CLINICAL TRIAL: NCT04680728
Title: Venous Congestion and Organ Dysfunction in Intensive Care: a Prospective, Multicenter, Observational Study to Evaluate Prevalence and Risk Factors.
Brief Title: Venous Congestion and Organ Dysfunction.
Acronym: CoDoRéa
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GUINOT 2020
Record Dates: First submitted 2020-11-23; First posted 2020-12-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Venous Congestion; Organ Dysfunction Syndrome
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: Patient admitted to intensive care for less than 24 hours.
  Interventions: Other: collection of biological parameters; Other: collection of echographic parameters; Other: collection of clinical parameters

INTERVENTIONS:
Other: collection of biological parameters — haemoglobin, haematocrit, sodium, chloraemia, total protein, albumin, L-lactate, pro-BNP, creatinine, uremia, AST, ALT, GGT, ALP, bilirubin, prothrombin time, urinary test if available.
Other: collection of echographic parameters — echocardiography (FEVG, subaortic ITV before and after LJP, cardiac index, MAPSE, mitral flow doppler, RVFAC, FEVD, STDVD, VD/VG ratio, TAPSE, tricuspid S wave, IT with PAPs, tricuspid flow doppler), Doppler of suprahepatic veins (S wave, D wave, S/D ratio), renal doppler (VII, RRI, aspect of venous flow in cortical and hilar), femoral venous doppler, doppler of the portal trunk, diameter of the VCI.
Other: collection of clinical parameters — eason for hospitalisation, co-morbidities, IGS2 score, SOFA, haemodynamic signs (BP, HR, CVP), sinus rhythm or not, temperature, diuresis, weight, input-output assessment, use of dialysis, ventilatory parameters (intubation, mode, FiO2(%), Vt, FR, PEEP, plateau pressure, driving pressure), state of shock (sepsis, postoperative, haemorrhagic, cardiogenic), transfusion (type, number), catecholamines (type, dose, duration), diuretics and dose, clinical criteria of venous congestion (jugular turgidity, hepato-jugular reflux, hepatosplenomegaly, pitting oedemas of the lower limbs, hepatalgia), neurological evaluation (Glasgow Coma Scale, CAM-ICU), time to resume enteral feeding and bowel movements, weight.

SUMMARY:
Venous congestion, which is a phenomenon described in cardiology and post-operative cardiac surgery, is responsible for an increase in morbidity and mortality.

Indeed, it can lead to kidney failure, liver failure, prolonged ileus, scarring complications, and neurological disorders. Clinical and ultrasound indications have been described to diagnose this condition.

To date, this phenomenon is poorly known and not described in intensive care patients outside the cardiac context. However, intensive care patients can present the risk factors associated with the occurrence of congestion: acute cardiac failure, significant water-salt overload, and/or fluid distribution anomalies. Thus, observational studies have found an association between the input-output balance, the quantity of salt-water intake, the presence of right heart dysfunction and the occurrence of acute kidney failure, digestive disorders, hypoxemia and a prolonged stay in intensive care. The presence of a congestive condition is medically treatable since diuretic decongestion is associated with improved cardiac outcomes.

It is therefore necessary, in an intensive care context, to be able to define and diagnose this state of venous congestion, to study its prevalence, and to confirm the existence of a link with organ failure in order to pave the way to known adapted treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Patient who has expressed his or her non-opposition to the collection of data (or the health care proxy, or a close relative if the patien is unable to receive the information)
* Patient admitted to intensive care for less than 24 hours.

Exclusion Criteria:

* Person not affiliated to the national health insurance
* Minor, protected major
* Pregnant or breastfeeding women
* Anechogenicity confirmed by the operator
* Chronic atrial fibrillation
* Mechanical cardiac assistance
* Uncontrolled blood pressure (MAP < 65 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient admitted to intensive care for less than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
the presence of venous congestion | From date of inclusion until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 28 day

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Andrei S, Bahr PA, Nguyen M, Bouhemad B, Guinot PG. Prevalence of systemic venous congestion assessed by Venous Excess Ultrasound Grading System (VExUS) and association with acute kidney injury in a general ICU cohort: a prospective multicentric study. Crit Care. 2023 Jun 8;27(1):224. doi: 10.1186/s13054-023-04524-4. PMID 37291662
- [Derived] Andrei S, Longrois D, Nguyen M, Bouhemad B, Guinot PG. Portal vein pulsatility is associated with the cumulative fluid balance: A post hoc longitudinal analysis of a prospective, general intensive care unit cohort. Eur J Anaesthesiol. 2025 Apr 1;42(4):324-331. doi: 10.1097/EJA.0000000000002111. Epub 2024 Dec 16. PMID 39686672
- [Derived] Guinot PG, Longrois D, Andrei S, Nguyen M, Bouhemad B; CodOrea study group. Exploring congestion endotypes and their distinct clinical outcomes among ICU patients: A post-hoc analysis. Anaesth Crit Care Pain Med. 2024 Jun;43(3):101370. doi: 10.1016/j.accpm.2024.101370. Epub 2024 Mar 8. PMID 38462160